CLINICAL TRIAL: NCT05248243
Title: Recruitment Assessment in Patients With Acute Respiratory Distress Syndrome and Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramos Mejía Hospital (Other)
Responsible Party: Principal Investigator, Roberto Santa Cruz, Principal Investigator, Ramos Mejía Hospital
Other Study IDs: Hospital General Ramos Mejía
Record Dates: First submitted 2022-02-15; First posted 2022-02-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19 Pneumonia; Recruitment
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Recruitment assessment — Intervention Details:
  Construction of the P/V curve with subsequent measurement of HR and Vmax.

SUMMARY:
Respiratory failure associated with Covid-19 can be expressed as acute respiratory distress syndrome (ARDS), which is an acute inflammatory lung injury,which generally requires the use of invasive mechanical ventilation (MV). There are inconclusive results regarding the potential lung recruitment in ARDS.

At the lung level, the relationship between lung volume and pressure can be graphed through a pressure/volume (P/V) curve. In this curve, hysteresis (H) can be evaluated, which is the amount of energy generated during inspiration that is not recovered during expiration. H is related to recruitment, assuming that the greater H the greater the alveolar recruitment. For this reason, the objective of this study is the measurement of H as a way to assess the lung recruitment capacity, in patients with ARDS and in patients with Covid-19 who develop ARDS (ARDS- Covid)

DETAILED DESCRIPTION:
During the first 7 days of the patient on mechanical ventilation (MV), measurements will be taken. For this, the patient will be in the supine position (DS) or the prone position (DP). The patient will be on a dose of analgesics, under sedation and muscle relaxation and will not present any respiratory stimulus.

Data from MV will also be recorded (prior to recruitment assessment): tidal volume (TV) in milliliters (ml), respiratory rate (RR) in a minute, fraction of inspired oxygen (FiO2), positive end-expiratory pressure (PEEP), in centimeters of water (cmH2O), plateau pressure (Pplat, measured after an end-inspiratory pause, cmH2O), mean airway pressure (PM, cmH2O), minute volume (calculated as the product of RR and TV) in milliliters per minute, ∆P (calculated as Pplat minus PEEP, cmH2O), static compliance (calculated as TV divided by ∆P, ml/cmH2O). Arterial blood gases will also be considered.

The proposed recruitment assessment will be the measurement of pulmonary hysteresis ratio. For measurements, a ventilator (Neumovent GraphNet Advance-TS, Córdoba Argentina) will be used. Additionally, a dedicated software connected to a computer will be used to perfThe evaluation of pressure in relation to volume will also be carried out, through the pressure/volume curve (PV curve), available in the respirator. A low-flow inflation and deflation PV curve from 0 up to 40 cm H2O and from 40 down to 0 cm H2O will be performed using the automatic tool on the ventilator (P/V tool; Neumovent GraphNet Advance-ts, Córdoba Argentina). The P-V curve can be visualized immediately on the screen of the mechanical ventilator and will be taken as a method to assess lung recruitment through the hysteresis-like behavior of the respiratory system. Inﬂation and deﬂation volume data will be corrected for changes in oxygen consumption.

Ratio hysteresis (RH) of the respiratory system will be measured by planimetry using SigmaPlot 12.0 software. There, through a cursor, for the measurement of hysteresis, the place where the volume was greater was drawn and the coincident pressure value was considered. Subsequently the ratio hysteresis will be calculated as the ratio between hysteresis and the product of the pressure span and the maximum volume reached (maximum hysteresis). Also, through the maximum distance between the inspiratory and expiratory limb of the curve weighted by the maximum volume, the normalized maximum distance (Vmax) is calculated. Recruitment potential will considered when there is a HR ≥ 28% and aVmax ≥ 41%.

Data Analysis. Categorical variables will be presented as number and percentage, while continuous variables will be presented as mean and standard deviation or median and interquartile range, as appropriate. The Chi2 test or Fisher's exact test will be used for qualitative variables and the Student test or the Mann-Whitney U test for quantitative variables. To evaluate correlation, the Pearson or Spearman test will be used, according to the distribution of the evaluated variables. A p ≤ 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have been receiving MV with diagnosis of ARDS (Berlin definition) and ARDS-Covid-19.

Exclusion Criteria:

* Patients with chronic pulmonary disease
* Patients with a high risk of death within 3 months for reasons other than ARDS-Covid-19
* Patients having made the decision to withhold life-sustaining treatment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 15 years of age or older who have been receiving MV in the first 7 days and have been defined as ARDS and ARDS-Covid-19 (with a positive polymerase chain reaction in nasopharyngeal swab samples) according to the clinical criteria of the Berlin definition.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Potential recruitment of patients with ARDS and ARDS-Covid-19 | First 7 days of the patient on mechanical ventilation (MV)
  Recruitment potential will considered when there is a HR ≥ 28% and Vmax ≥ 41%.

SECONDARY OUTCOMES:
Assess the association between APACHE II (Acute Physiology And Chronic Health Evaluation) score and and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between APACHE and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
  Tidal volume and pressure will be combined to report the Recruitment Index (R/I) in mL/cmH2O.
  A threshold of 0.5 will be used to deﬁne high recruitability (R/I ratio >= 0.5 ml/cmH2O) and low recruitability (R/I ratio < 0.5 ml/cmH2O).
Assess the association between TV and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between TV and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between plateau pressure and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between plateau pressure and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
  * Oxygenation: PaO2/FiO2 (ratio between arterial oxygen pressure and inspired fraction of oxygen).
  * Static compliance (cmH2O)
  * Plateau pressure (cmH2O)
  * ∆P (ml/cmH2O)
  Tidal volume and pressure will be combined to report the Recruitment Index (R/I) in mL/cmH2O.
Assess the association between ΔP and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between ΔP and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between static compliance and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between static compliance and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between mechanical power and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between mechanical power and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between PaO2/FiO2 and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between PaO2/FiO2 and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between PaCO2 and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between PaCO2 and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).
Assess the association between ventilator free days (in days) and potential recruitment | First 7 days of the patient on mechanical ventilation (MV)
  Assess the correlation between ventilator free days (in days) and potential recruitment (HR ≥ 28% and Vmax ≥ 41%).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Agudos Ramos Mejía, Ciudad Autonoma de Buenos Aire, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Ziehr DR, Alladina J, Petri CR, Maley JH, Moskowitz A, Medoff BD, Hibbert KA, Thompson BT, Hardin CC. Respiratory Pathophysiology of Mechanically Ventilated Patients with COVID-19: A Cohort Study. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1560-1564. doi: 10.1164/rccm.202004-1163LE. No abstract available. PMID 32348678
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Chiumello D, Arnal JM, Umbrello M, Cammaroto A, Formenti P, Mistraletti G, Bolgiaghi L, Gotti M, Novotni D, Reidt S, Froio S, Coppola S. Hysteresis and Lung Recruitment in Acute Respiratory Distress Syndrome Patients: A CT Scan Study. Crit Care Med. 2020 Oct;48(10):1494-1502. doi: 10.1097/CCM.0000000000004518. PMID 32897667
- [Result] Demory D, Arnal JM, Wysocki M, Donati S, Granier I, Corno G, Durand-Gasselin J. Recruitability of the lung estimated by the pressure volume curve hysteresis in ARDS patients. Intensive Care Med. 2008 Nov;34(11):2019-25. doi: 10.1007/s00134-008-1167-8. Epub 2008 Jun 25. PMID 18575846
- [Result] Chen L, Del Sorbo L, Grieco DL, Shklar O, Junhasavasdikul D, Telias I, Fan E, Brochard L. Airway Closure in Acute Respiratory Distress Syndrome: An Underestimated and Misinterpreted Phenomenon. Am J Respir Crit Care Med. 2018 Jan 1;197(1):132-136. doi: 10.1164/rccm.201702-0388LE. No abstract available. PMID 28557528
- [Result] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Result] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Derived] Hohmann F, Wedekind L, Grundeis F, Dickel S, Frank J, Golinski M, Griesel M, Grimm C, Herchenhahn C, Kramer A, Metzendorf MI, Moerer O, Olbrich N, Thieme V, Vieler A, Fichtner F, Burns J, Laudi S. Early spontaneous breathing for acute respiratory distress syndrome in individuals with COVID-19. Cochrane Database Syst Rev. 2022 Jun 29;6(6):CD015077. doi: 10.1002/14651858.CD015077. PMID 35767435